CLINICAL TRIAL: NCT01988922
Title: Role of CYP2B6 Polymorphisms in Ketamine Metabolism and Clearance
Brief Title: CYP2B6 Polymorphisms in Ketamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201307034
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers
Keywords: ketamine polymorphisms
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine arm- *1/*1 (Experimental): 1.*1/*1- oral racemic ketamine 0.4 mg/kg
  Interventions: Drug: ketamine
- Ketamine arm - *1/*6 (Experimental): 2. *1/*6- oral racemic ketamine 0.4 mg/kg
  Interventions: Drug: ketamine
- Ketamine arm - *6/*6 (Experimental): 3. *6/*6- oral racemic ketamine 0.4 mg/kg
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — 0.4 mg/kg oral racemic ketamine

SUMMARY:
This research study will determine if genetic variation in CYP2B6 affects how the body metabolizes ketamine.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 yr old
2. CYP2B6*1/*1, CYP2B6*1/*6 or CYP2B6*6/*6 genotype (see table) (Note: subjects of other rare genotype but with one or more 516G>T, 785A>G, 983T>C or 1459C>T polymorphism may be enrolled at PI's discretion)
3. Good general health with no remarkable medical conditions
4. BMI <33
5. Provided informed consent

Exclusion Criteria:

1. Known history of liver or kidney disease
2. Use of prescription or non prescription medications, herbals, foods or chemicals known to be metabolized by or affecting CYP2B6
3. Females who are pregnant or nursing
4. Known history of drug or alcohol addiction (prior or present addiction or treatment for addiction)
5. Direct physical access to and routine handling of addicting drugs in the regular course of duty (this is a routine exclusion from studies of drugs with addiction potential)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Rao, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Arm- *1/*1: 1.*1/*1- oral racemic ketamine 0.4 mg/kg
  ketamine: 0.4 mg/kg oral racemic ketamine as a one-time dose
- Ketamine Arm - *1/*6: 2. *1/*6- oral racemic ketamine 0.4 mg/kg
  ketamine: 0.4 mg/kg oral racemic ketamine as a one-time dose
- Ketamine Arm - *6/*6: 3. *6/*6- oral racemic ketamine 0.4 mg/kg
  ketamine: 0.4 mg/kg oral racemic ketamine as a one-time dose
Period: Overall Study
Arm/Group | Ketamine Arm- *1/*1 | Ketamine Arm - *1/*6 | Ketamine Arm - *6/*6
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Arm- *1/*1 | Ketamine Arm - *1/*6 | Ketamine Arm - *6/*6 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6) | 27 (11) | 37 (13) | 29 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 7 | 6 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Effects of CYP2B6 Genetic Variants on Ketamine Metabolism and Clearance by CYP2B6*6 Hetero or Homozygote Genotype.
Description: Ketamine metabolism, measured as the plasma norketamine/ketamine AUC ratio in CYP2B6*6 carriers (CYP2B6*6 hetero or homozygotes) compared to the wild-type CYP2B6*1/*1 genotype Ketamine, norketamine, and dehydronorketamine concentrations in plasma and urine were determined by enantioselective HPLC tandem mass spectrometry, using solid phase extraction, based on a modification of a published method.
Time Frame: up to 24 hours
Population: 3 genotype groups, metabolism measured for both R- and S-ketamine
Measure: Mean (Standard Deviation); unit: ng/ml*hr
Arm/Group | R-ketamine *1/*1 | S-ketamine *1/*1 | R-ketamine *1/*6 | S-ketamine *1/*6 | R-ketamine *6/*6 | S-ketamine *6/*6
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ng/ml*hr | 29 (10) | 21 (7) | 26 (11) | 19 (10) | 35 (21) | 23 (13)
Statistical Analysis 1: Comparison: R-ketamine *1/*1 vs S-ketamine *1/*1 vs R-ketamine *1/*6 vs S-ketamine *1/*6 vs R-ketamine *6/*6 vs S-ketamine *6/*6; Test type: Other — Differences between CYP2B6*1/*1, CYP2B6*1/*6, and CYP2B6*6/*6 genotypes for pharmacokinetic parameters were analyzed using one-way ANOVA followed by the Student-Newman-Keuls test for multiple comparisons (Sigmaplot 12.5; Systat Software, Inc, USA). Nonnormal data were log transformed for analysis but reported as the nontransformed results; p < 0.05, ANOVA; One-way ANOVA followed by the Student-Newman-Keuls test for multiple comparisons

ADVERSE EVENTS:
Arm/Group | Ketamine Arm- *1/*1 | Ketamine Arm - *1/*6 | Ketamine Arm - *6/*6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2013-07-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT01988922/Prot_000.pdf
  • Statistical Analysis Plan (2013-07-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT01988922/SAP_001.pdf